CLINICAL TRIAL: NCT03367663
Title: The Effect of Prednisone on Atherogenesis as Studied in the Macrophage Foam Cell Formation Model System.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Prof. Tony hayek MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Tony hayek MD, Director, Department of Internal Medicine E, Rambam Health Care Campus
Organization: Rambam Health Care Campus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0254-17-RMB
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Atherosclerosis; Dyslipidemias; Diabetes
MeSH Terms: conditions — Atherosclerosis; Dyslipidemias; Diabetes Mellitus | interventions — Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low dose (Experimental): Each participant will be randomly assigned to one of two treatment groups, low dose of Prednisone 20mg/d (n=10) and high dose of Prednisone 40 mg/d (n=10). During the experimental periods, the subjects will take either one or two 20mg tablet of Prednisone, according to their assigned group. Subjects will be instructed to take the tablets at home in the mornings after a meal each day for 5 consecutive days. At the baseline visit, a medical history will be documented and a physical examination will be performed. Subjects will be asked to come to the research unit on days 1,2,5 after a 14h fasting where two blood samples (5ml each) will be taken, immediately centrifuged, one for biochemical analysis (Lipid profile, Liver function tests, Glucose, Electrolytes and Renal function tests) and the second will be aliquoted, and stored at -20°C until later analyses.
  Interventions: Drug: Prednisone 20 Mg
- high dose (Experimental): Each participant will be randomly assigned to one of two treatment groups, low dose of Prednisone 20mg/d (n=10) and high dose of Prednisone 40 mg/d (n=10). During the experimental periods, the subjects will take either one or two 20mg tablet of Prednisone, according to their assigned group. Subjects will be instructed to take the tablets at home in the mornings after a meal each day for 5 consecutive days. At the baseline visit, a medical history will be documented and a physical examination will be performed. Subjects will be asked to come to the research unit on days 1,2,5 after a 14h fasting where two blood samples (5ml each) will be taken, immediately centrifuged, one for biochemical analysis (Lipid profile, Liver function tests, Glucose, Electrolytes and Renal function tests) and the second will be aliquoted, and stored at -20°C until later analyses.
  Interventions: Drug: Prednisone 40 Mg

INTERVENTIONS:
Drug: Prednisone 20 Mg — Each participant will be randomly assigned to one of two treatment groups, low dose of Prednisone 20mg/d (n=10) and high dose of Prednisone 40 mg/d (n=10). During the experimental periods, the subjects will take either one or two 20mg tablet of Prednisone, according to their assigned group. Subjects will be instructed to take the tablets at home in the mornings after a meal each day for 5 consecutive days. At the baseline visit, a medical history will be documented and a physical examination will be performed. Subjects will be asked to come to the research unit on days 1,2,5 after a 14h fasting where two blood samples (5ml each) will be taken, immediately centrifuged, one for biochemical analysis (Lipid profile, Liver function tests, Glucose, Electrolytes and Renal function tests) and the second will be aliquoted, and stored at -20°C until later analyses.
  Arms: low dose
Drug: Prednisone 40 Mg — Each participant will be randomly assigned to one of two treatment groups, low dose of Prednisone 20mg/d (n=10) and high dose of Prednisone 40 mg/d (n=10). During the experimental periods, the subjects will take either one or two 20mg tablet of Prednisone, according to their assigned group. Subjects will be instructed to take the tablets at home in the mornings after a meal each day for 5 consecutive days. At the baseline visit, a medical history will be documented and a physical examination will be performed. Subjects will be asked to come to the research unit on days 1,2,5 after a 14h fasting where two blood samples (5ml each) will be taken, immediately centrifuged, one for biochemical analysis (Lipid profile, Liver function tests, Glucose, Electrolytes and Renal function tests) and the second will be aliquoted, and stored at -20°C until later analyses.
  Arms: high dose

SUMMARY:
Glucocorticoids (GCs) are a class of endogenous steroid hormones produced by the adrenal glands and controlled by the hypothalamic-pituitary-adrenal axis (HPA). One of the mechanisms of their action is achieved through ligand-receptor attachment to a class of cytosolic steroid hormone receptors termed Glucocorticoid Receptors (GRs). The formed ligand-receptor complex is a transcription factor involved in gene activation of anti-inflammatory products or repression of pro-inflammatory products [1]. Synthetic forms of GCs are a group of anti-inflammatory and immunosuppressive medications (e.g. Prednisone) that are widely used in clinical practice to treat inflammatory diseases (e.g. Rheumatoid Arthritis, Vasculitis, Asthma). The effectiveness of this class of drugs is limited by numerous adverse effects that include, but not limited to, insulin resistance, glucose intolerance, dyslipidemia, and hypertension, all of which are well known risk factors for cardiovascular diseases (CVD) [2,3]. Furthermore, recent research suggest that inflammation has a key role in development of CVD and can predict prognosis [4]. Inflammatory cells have an important role in the development of atherosclerotic lesion in the arteries. Blood monocyte-derived macrophages are involved in this process, and they infiltrate the lesion where they take up various forms of lipids (cholesterol - rich LDL, and oxidized LDL) as well as triglycerides - rich VLDL), followed by the formation of lipid-laden foam cells, the hallmark of early atherogenesis. Inflammatory cells and molecules as well as proteolytic enzymes secreted from inflammatory cells in the atherosclerotic lesion, have a central role in destabilizing the plaque (vulnerable plaque) leading to its rupture, which, in turn, induces thrombosis, and initiating acute coronary events [4,5].

Based on our understanding of the involvement of inflammation in the early development of atherosclerotic lesion, and our experience with the anti-inflammatory effects of synthetic GCs, a hypothesis emerged suggesting this class of drugs as a way to inhibit early atherosclerotic plaque formation, and to attenuate CVDs [6]. Research results in this field are surprising because while glucocorticoids treatment in humans increase the risk of CVDs [6,7,8,9], animal models shows the opposite, atheroprotection was shown in rabbits [10,11,12] and mice [13,14,15]. This paradox may be explained partially by the fact that clinical studies in this field are mainly conducted in patients with predisposing factors to develop CVD, either because of pre-existing traditional risk factors like Diabetes and Hyperlipidemia, or because of the pre-existing medical condition they are being treated for with GCs (e.g. Rheumatoid Arthritis). Mechanism based research to study the effects of GCs on atherogenesis, without confounding factors, is lacking. Only few studies were performed on GCs in healthy subjects but none of them explored their effects on foam cell formation [16,17].

Our study thus aims to further our understanding of the role of specific glucocorticoid, prednisone, in the process of atherogenesis. In order to achieve that we plan to study the following: 1. The effects of five days of treatment with prednisone on serum lipid concentration and oxidative stress. 2. an Ex-vivo study is planned where the serum of healthy human subjects treated with Prednisone, will be introduced to J774A.1 murine macrophage-like cell line, a well-studied macrophage foam cell formation model.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between the ages of 18-50 years of age, with a body mass index within the range of 18 to 27 kg/m2, with no previous medical history of illnesses or drug allergy and with no current medical treatments.

Exclusion Criteria:

* Students or hospital employees under the direct supervision of the PI or lead researcher. Any previous history of acute or chronic illnesses including but not limited to Cardiovascular, Pulmonary, Gastrointestinal, Renal, Endocrinal, Cancer, Diabetes or Pre-Diabetes (HbA1c > 5.5%), Hypertension, Dyslipidemia, Smoking, or who had taken glucocorticoids within the previous 3 months before the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2018-07-09 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Serum atherogenicity | 3 months
  Macrophage lipids (triglycerides and cholesterol) content (μg/mg cell protein) following incubation with serum derived from the subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Hayek, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cohen DM, Steger DJ. Nuclear Receptor Function through Genomics: Lessons from the Glucocorticoid Receptor. Trends Endocrinol Metab. 2017 Jul;28(7):531-540. doi: 10.1016/j.tem.2017.04.001. Epub 2017 May 8. PMID 28495406
- [Background] Stahn C, Buttgereit F. Genomic and nongenomic effects of glucocorticoids. Nat Clin Pract Rheumatol. 2008 Oct;4(10):525-33. doi: 10.1038/ncprheum0898. Epub 2008 Sep 2. PMID 18762788
- [Background] Schacke H, Docke WD, Asadullah K. Mechanisms involved in the side effects of glucocorticoids. Pharmacol Ther. 2002 Oct;96(1):23-43. doi: 10.1016/s0163-7258(02)00297-8. PMID 12441176
- [Background] Hansson GK. Inflammation, atherosclerosis, and coronary artery disease. N Engl J Med. 2005 Apr 21;352(16):1685-95. doi: 10.1056/NEJMra043430. No abstract available. PMID 15843671
- [Background] Dickhout JG, Basseri S, Austin RC. Macrophage function and its impact on atherosclerotic lesion composition, progression, and stability: the good, the bad, and the ugly. Arterioscler Thromb Vasc Biol. 2008 Aug;28(8):1413-5. doi: 10.1161/ATVBAHA.108.169144. No abstract available. PMID 18650503
- [Background] Walker BR. Glucocorticoids and cardiovascular disease. Eur J Endocrinol. 2007 Nov;157(5):545-59. doi: 10.1530/EJE-07-0455. PMID 17984234
- [Background] del Rincon I, O'Leary DH, Haas RW, Escalante A. Effect of glucocorticoids on the arteries in rheumatoid arthritis. Arthritis Rheum. 2004 Dec;50(12):3813-22. doi: 10.1002/art.20661. PMID 15593231
- [Background] del Rincon I, Battafarano DF, Restrepo JF, Erikson JM, Escalante A. Glucocorticoid dose thresholds associated with all-cause and cardiovascular mortality in rheumatoid arthritis. Arthritis Rheumatol. 2014 Feb;66(2):264-72. doi: 10.1002/art.38210. PMID 24504798
- [Background] Ajeganova S, Svensson B, Hafstrom I; BARFOT Study Group. Low-dose prednisolone treatment of early rheumatoid arthritis and late cardiovascular outcome and survival: 10-year follow-up of a 2-year randomised trial. BMJ Open. 2014 Apr 7;4(4):e004259. doi: 10.1136/bmjopen-2013-004259. PMID 24710131
- [Background] Cavallero C, Di Tondo U, Mingazzini PL, Nicosia R, Pericoli MN, Sarti P, Spagnoli LG, Villaschi S. Cell proliferation in the atherosclerotic plaques of cholesterol-fed rabbits. Part 3. Histological and radioautographic observations on glucocorticoids-treated rabbits. Atherosclerosis. 1976 Nov-Dec;25(2-3):145-52. doi: 10.1016/0021-9150(76)90020-4. PMID 1008903
- [Background] Makheja AN, Bloom S, Muesing R, Simon T, Bailey JM. Anti-inflammatory drugs in experimental atherosclerosis. 7. Spontaneous atherosclerosis in WHHL rabbits and inhibition by cortisone acetate. Atherosclerosis. 1989 Apr;76(2-3):155-61. doi: 10.1016/0021-9150(89)90099-3. PMID 2543422
- [Background] Asai K, Funaki C, Hayashi T, Yamada K, Naito M, Kuzuya M, Yoshida F, Yoshimine N, Kuzuya F. Dexamethasone-induced suppression of aortic atherosclerosis in cholesterol-fed rabbits. Possible mechanisms. Arterioscler Thromb. 1993 Jun;13(6):892-9. doi: 10.1161/01.atv.13.6.892. PMID 8499410
- [Background] Auvinen HE, Wang Y, Princen H, Romijn JA, Havekes LM, Smit JW, Meijer OC, Biermasz NR, Rensen PC, Pereira AM. Both transient and continuous corticosterone excess inhibit atherosclerotic plaque formation in APOE*3-leiden.CETP mice. PLoS One. 2013 May 22;8(5):e63882. doi: 10.1371/journal.pone.0063882. Print 2013. PMID 23717502
- [Background] Out C, Dikkers A, Laskewitz A, Boverhof R, van der Ley C, Kema IP, Wolters H, Havinga R, Verkade HJ, Kuipers F, Tietge UJ, Groen AK. Prednisolone increases enterohepatic cycling of bile acids by induction of Asbt and promotes reverse cholesterol transport. J Hepatol. 2014 Aug;61(2):351-7. doi: 10.1016/j.jhep.2014.03.025. Epub 2014 Mar 26. PMID 24681341
- [Background] Tauchi Y, Zushida L, Chono S, Sato J, Ito K, Morimoto K. Effect of dexamethasone palmitate-low density lipoprotein complex on cholesterol ester accumulation in aorta of atherogenic model mice. Biol Pharm Bull. 2001 Aug;24(8):925-9. doi: 10.1248/bpb.24.925. PMID 11510487
- [Background] Fleishaker DL, Mukherjee A, Whaley FS, Daniel S, Zeiher BG. Safety and pharmacodynamic dose response of short-term prednisone in healthy adult subjects: a dose ranging, randomized, placebo-controlled, crossover study. BMC Musculoskelet Disord. 2016 Jul 16;17:293. doi: 10.1186/s12891-016-1135-3. PMID 27424036
- [Background] Kauh EA, Mixson LA, Shankar S, McCarthy J, Maridakis V, Morrow L, Heinemann L, Ruddy MK, Herman GA, Kelley DE, Hompesch M. Short-term metabolic effects of prednisone administration in healthy subjects. Diabetes Obes Metab. 2011 Nov;13(11):1001-7. doi: 10.1111/j.1463-1326.2011.01432.x. PMID 21635675
- [Background] Nikitina NA, Sobenin IA, Myasoedova VA, Korennaya VV, Mel'nichenko AA, Khalilov EM, Orekhov AN. Antiatherogenic effect of grape flavonoids in an ex vivo model. Bull Exp Biol Med. 2006 Jun;141(6):712-5. doi: 10.1007/s10517-006-0260-7. English, Russian. PMID 17364057
- [Background] Hamoud S, Hayek T, Volkova N, Attias J, Moscoviz D, Rosenblat M, Aviram M. Pomegranate extract (POMx) decreases the atherogenicity of serum and of human monocyte-derived macrophages (HMDM) in simvastatin-treated hypercholesterolemic patients: a double-blinded, placebo-controlled, randomized, prospective pilot study. Atherosclerosis. 2014 Jan;232(1):204-10. doi: 10.1016/j.atherosclerosis.2013.11.037. Epub 2013 Nov 19. PMID 24401239